CLINICAL TRIAL: NCT01473238
Title: Desktop vs. Mobile Data Collection in a Prospective Multicenter Clinical Trial
Brief Title: Desktop Versus Mobile Data Collection in Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PSP_Appendix_2
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: User Experience
Keywords: Desktop computer; Mobile; iPad; Evaluation; User experience; Benefits; Cost analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desktop PC (Active Comparator): Conventional institutional Desktop Personal Computers will be used to collect data of patients via a password protected encrypted interface.
  Interventions: Other: Evaluation form
- Mobile (Experimental): Novel Mobile Clinical Trial Management System on iPads will be used to collect data of patients via a password protected encrypted interface.
  Interventions: Other: Evaluation form

INTERVENTIONS:
Other: Evaluation form — A validated user experience evaluation questionnaire will be completed by each participant in the beginning, at the interim period, and at the end of the trial
  Other Names: User evaluation questionnaire; User experience form

SUMMARY:
Paper-based data collection for prospective clinical trials is associated with a poor quality of data collection. This typically involves missing or wrong data entry or a low recruitment rate, mainly due to the cumbersome and uncontrolled data collection.

Electronic data collection is associated with improved quality of data entry in the cases of Electronic Patient Records (EPR) and patient handover among doctors during night and day shifts. However, a comprehensive direct comparison between web-based desktop personal computer (PC) and mobile (e.g. iPad) data collection has not yet been reported.

The purpose of this prospective trial is to compare the users' experience with the web-based desktop PC and mobile data collection (iPad) tools.

DETAILED DESCRIPTION:
The investigators designed a prospective randomized controlled trial where doctors from several randomly selected hospitals will use either a desktop PC or mobile (iPad) data collection tool. A validated user experience evaluation instrument will be used at the beginning, during interim analysis and at the end of the trial.

The desktop-based data collection is built on Drupal, a renowned open source content management system (CMS). The same CMS will be used with a special interface designed for iOS/iPad. Both data collection platforms will be used in parallel to a prospective clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Room doctors
* Surgeons
* Agree to participate in the trial
* Provide informed consent
* Have basic information technology literacy
* Agree to receive brief training of the platform

Exclusion Criteria:

* Clinicians and health care professionals not part of this trial
* Lacking of basic information technology literacy

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation score | 2 years
  A validated user experience and evaluation instrument will be used.
  The overall score will be compared between the Desktop PC and Mobile (iPad) data collection tools.
  PC: indicates Personal Computer

SECONDARY OUTCOMES:
Recruitment rate | 2 years
  The recruitment rate is defined as the proportion of patients recruited divided by the total number of patients recruited + patients missed: (rate=recruited/(recruited+missed).
  The recruitment rates will be compared between the Desktop PC and Mobile (iPad) data collection tools.
  PC: indicates Personal Computer
Cost-effectiveness analysis | 2 years
  Cost-effectiveness analysis (CEA) is a form of economic analysis that compares the relative costs and outcomes (effects) of two or more courses of action. CEA assigns a monetary value to the measure of effect. Typically the CEA is expressed in terms of a ratio where the denominator is a gain from a measure and the numerator is the cost associated with this gain.
  In this study, CEA will be calculated as: (ratio=costs/evaluation score) and (ratio=costs/recruitment rate).
Cost-benefit analysis | 2 years
  Cost-benefit analysis (CBA) is a systematic process for calculating and comparing benefits and costs of a project for two purposes; in order to determine if it is a sound investment (justification/feasibility), and to see how it compares with alternate projects (ranking/priority assignment). It involves comparing the total expected cost of each option against the total expected benefits, to see whether the benefits outweigh the costs, and by how much. In CBA, benefits and costs are expressed in money terms, and are adjusted for the "time value of money".
Cost-utility analysis | 2 years
  Cost-utility analysis (CUA) is a form of financial analysis used to guide procurement decisions. The most common and well-known application of this analysis is in health technology assessment. Cost is measured in monetary units.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri A Raptis, MD, MSc, Principal Investigator — University Hospital Zurich, Department of Surgery; Rolf Graf, PhD, Principal Investigator — University Hospital Zurich, Department of Surgical Research
Locations (2):
- Switzerland (2):
  - University of St. Gallen, Institute of Information Managemen, Sankt Gallen
  - University Hospital Zurich, Department of Surgery, Zurich

REFERENCES:
- [Background] Raptis DA, Mettler T, Tzanas K, Graf R. A novel open-source web-based platform promoting collaboration of healthcare professionals and biostatisticians: a design science approach. Inform Health Soc Care. 2012 Jan;37(1):22-36. doi: 10.3109/17538157.2011.590257. Epub 2011 Oct 19. PMID 22010822
- [Background] Raptis DA, Fernandes C, Chua W, Boulos PB. Electronic software significantly improves quality of handover in a London teaching hospital. Health Informatics J. 2009 Sep;15(3):191-8. doi: 10.1177/1460458209337431. PMID 19713394
- [Background] Mirani R, Lederer A. An Instrument for Assessing the Organizational Benefits of IS projects. Decision Sciences, Vol. 29, No. 4, 1998, 803-838.
- See also: An Instrument for Assessing the Organizational Benefits of IS Projects — http://onlinelibrary.wiley.com/doi/10.1111/j.1540-5915.1998.tb00878.x/abstract